CLINICAL TRIAL: NCT04290351
Title: Comparative Study of Band Ligation and Phlebotonic Drug Versus Only Phlebotonic Drug, in Bleeding Internal Hemorrhoids.
Brief Title: The Effect of Rubber Band Ligation in Bleeding Internal Hemorrhoids.
Status: Completed | Type: Observational
Sponsor: Konya Meram State Hospital (Other)
Responsible Party: Principal Investigator, Alpaslan Şahin, principal investigators, Konya Meram State Hospital
Other Study IDs: hemorrhoids X. study
Record Dates: First submitted 2020-02-25; First posted 2020-02-28 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Hemorrhoids, Internal
MeSH Terms: conditions — Hemorrhoids

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Band ligation and phlebotonic group: Patients with rubber band ligation and the prescribed anti hemorrhoidal drug will be examined in this group.
  (Note: The researcher has no contribution or intervention to the treatment method.)
  Interventions: Procedure: band ligation; Drug: oral 450 mg diosmin+50 mg hesperidin
- Only phlebotonic group: Patients who are prescribed the only 450mg of diosmin + 50mg of hesperidin as a treatment for bleeding internal hemorrhoids will be examined in this group.
  (Note: The researcher has no contribution or intervention to the treatment method.)
  Interventions: Drug: oral 450 mg diosmin+50 mg hesperidin

INTERVENTIONS:
Procedure: band ligation — Rubber band ligation will be applied to patients, and then phlebotonic will be prescribed.
  (Note: The researcher has no contribution or intervention to the treatment method. Patients receiving this treatment will be observed.)
  Groups: Band ligation and phlebotonic group
Drug: oral 450 mg diosmin+50 mg hesperidin — 450 mg diosmin + 50 mg hesperidin will be prescribed to patients undergoing band ligation.
  (Note: The researcher has no contribution or intervention to the treatment method. Patients receiving this treatment will be observed.)

SUMMARY:
In this study, the researchers planned to compare the treatment results of patients undergoing rubber band ligation in addition to drug therapy in hemorrhagic internal hemorrhoids patients and those treated only with anti-hemorrhoidal drugs.

DETAILED DESCRIPTION:
Introduction: Band ligation is one of the most frequently used methods in the treatment of hemorrhagic internal hemorrhoidal disease. Also, phlebotonic use and surgical excision options are available as an anti-hemorrhoidal drug in the treatment of the disease. Many studies have shown that these methods are safe to use. Band ligation is used quite often in our clinic. Whether or not band ligation is performed, these patients are prescribed phlebotonics as an anti-hemorrhoidal drug.

Purpose: In this study, investigators aimed to investigate the benefit of adding rubber band ligation to treatment in hemorrhagic internal hemorrhoidal disease treated with the anti hemorrhoidal drug.

Method: The study was planned prospectively and observationally. Patients are not assigned to groups by the researcher. The researcher cannot interfere with the treatment method given to the patient. The method of treatment is the method approved by the patient's doctor.

Patients diagnosed with internal hemorrhoids will be examined in a group of patients who are prescribed anti-hemorrhoidal drugs and rubber band ligation in the context of routine treatment.

In the other group, again, in the form of routine treatment, patients who are not given rubber band ligation and who are given only anti-hemorrhoidal drugs will be examined.

Group 1: Patients who have been prescribed 450 mg diosmin + 50 mg hesperidin as an anti-hemorrhoidal drug and rubber band ligation will be included in this group.

Group 2: Patients who have been prescribed only 450 mg of diosmin + 50 mg of hesperidin as treatment, without rubber band ligation will be included in this group.

Patients will undergo a control examination in the 21 days after treatment.

* Whether the bleeding continues?
* Which bleeding day stopped?
* The comfort of the anal area will be evaluated
* Did the side effect develop?
* Did any complications occur? The above information will be entered into the SPSS program, and statistical analysis will be done.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with internal hemorrhoids with an anamnesis + examination + rectoscope.

Exclusion Criteria:

* Patients under 18 years old
* Patients over 65 years old
* Pregnant
* Chronic liver patients
* Those with bleeding disorders
* Patients taking anti-coagulants and anti-aggregates
* Patients with colorectal cancer.
* Those who have had hemorrhoid surgery before

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients between the ages of 18 and 65 who apply to our hospital from Konya and neighboring provinces and accept the treatments offered, constitute the study population.
Sampling Method: Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-12-20 (Actual)

PRIMARY OUTCOMES:
hemostasis rate | 21 days
  At the end of the treatment, the proportion of patients without hemorrhoids bleeding will be calculated.
Hemorrhage stopped on the day of treatment. | 21 days
  It will be determined that the bleeding stops on the day of treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Konya Training and Research Hospital, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lohsiriwat V. Treatment of hemorrhoids: A coloproctologist's view. World J Gastroenterol. 2015 Aug 21;21(31):9245-52. doi: 10.3748/wjg.v21.i31.9245. PMID 26309351
- [Background] Albuquerque A. Rubber band ligation of hemorrhoids: A guide for complications. World J Gastrointest Surg. 2016 Sep 27;8(9):614-620. doi: 10.4240/wjgs.v8.i9.614. PMID 27721924
- [Background] Schleinstein HP, Averbach M, Averbach P, Correa PAFP, Popoutchi P, Rossini LGB. ENDOSCOPIC BAND LIGATION FOR THE TREATMENT OF HEMORRHOIDAL DISEASE. Arq Gastroenterol. 2019 May 20;56(1):22-27. doi: 10.1590/S0004-2803.201900000-15. PMID 31141063